CLINICAL TRIAL: NCT02998749
Title: Agonal Breathing is a Positive Predictive Factor of Long Term Survival After Out-of-hospital Cardiac Arrest
Brief Title: Gasping Improves Long-term Survival After Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jiri Malek, Assoc. Prof.. MD, Ph.D., Charles University, Czech Republic
Other Study IDs: Gasping1
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Cardiac Arrest With Successful Resuscitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of our retrospective clinical study was to examine the association between agonal breathing, return of spontaneous circulation (ROSC), and long-term survival. A secondary aim was to examine role of basic life support (BLS) and response time. Our hypothesis is that agonal breathing has positive effects on both primary and secondary endpoints.

DETAILED DESCRIPTION:
Aims Agonal breathing ("gasping for air") has previously been found to be associated with the outcomes of out-of-hospital cardiac arrest (OHCA) patients on which resuscitation was attempted. On the other hand, little is known, about agonal breathing with regard to whether it is a positive factor for survival after hospital admission and how it relates to the patient's future quality of life. For this reason we have undertaken a retrospective study using a comprehensive emergency medical service (EMS) database from the Central Bohemian region of the Czech Republic. The primary endpoint of the study was to assess if agonal breathing present when EMS arrives has a positive impact on the six-month survival of OHCA patients, which was independent of other factors like EMS response time and BLS provision. The secondary endpoints sought to determine if agonal breathing positively impacts ROSC and an evaluation of various factors that can influence agonal breathing, specifically response time and provision of BLS.

Method The data were recorded using the Utstein protocol. Only anonymized data were used for analysis. The data were derived from the EMS registry of the Central Bohemian Region, which is the largest EMS in the Czech Republic. The study sample included all OHCA cases, of presumed cardiac origin, that where resuscitated by the EMS between 1st July 2013 and 30th June 2014 (n = 584). Two subsequent patient outcomes: (1) return of spontaneous circulation (defined as spontaneous circulation at hospital admission) and (2) six-month survival were assessed in patients with and without agonal breathing. Six-month survival data of OHCA patients of presumed cardiac origin was derived from administrative insurance registries or medical records of patients, with only aggregated data being available.

Factors that may influence the presence of agonal breathing, specifically BLS provision before a professional EMS team reached the patient and second, EMS team response times, were also examined. BLS provision by lay persons was reported by the first-on-scene EMS team as (yes/no) and phone assisted CPR was registered by the dispatcher as (yes/no). BLS was considered to have been provided if any of the following activities (1) resuscitation by a bystander, (2) phone assisted CPR, or (3) both were recorded as having been performed. The response time was calculated as the elapsed time between recorded activation of an EMS team and the on scene arrival time.

Other covariates such as age and sex were also available and analyzed. The initial difference in response time between the groups was assessed using the T-test. For categorical variables, the chi-square test was used. Simple and multivariate logistic regression models were used to assess relationships between factors related to the presence of agonal breathing and ROSC. A p-value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: all out-of-hospital cardiac arrest cases, of presumed cardiac origin, that where resuscitated by the emergency medical service of Central Bohemia region between 1st July 2013 and 30th June 2014 (n = 584) -

Exclusion Criteria: other than non-cardiac cause of cardiac arrest

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Victims of primary out-of-hospital cardiac arrest
Sampling Method: Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
association between agonal breathing and long-term survival | 6 months after successful resuscitation

SECONDARY OUTCOMES:
impact of agonal breathing on return of spontaneous circulation | immediately after resuscitation

IPD SHARING:
Plan to Share IPD: No